CLINICAL TRIAL: NCT05327439
Title: Using Alternative Nicotine Delivery Systems (ANDS) to Reduce Harm for Low SES Cigarette Smokers. (Tri-PEC Study)
Brief Title: Using ANDS to Reduce Harm for Low SES Cigarette Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2105002986
Record Dates: First submitted 2021-08-27; First posted 2022-04-14 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Smoking, Cigarette; Nicotine Dependence
Keywords: cigarette substitution; electronic nicotine delivery systems; ENDS; e-cigarette; nicotine pouch; nicotine dependence; low SES; smoking
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder; Vaping; Smoking | interventions — Nicotine; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Electronic Cigarette (Experimental): Participants in this experimental condition will be provided with a 4th generation electronic cigarette device and disposable cartridges.
  Interventions: Other: Nicotine (electronic cigarette)
- Nicotine Pouch (Experimental): Participants in this experimental condition will be provided with nicotine pouches.
  Interventions: Other: Nicotine (nicotine pouch)
- Smoking As Usual (No Intervention): Participants in this assessment-only condition will continue smoking as usual.

INTERVENTIONS:
Other: Nicotine (electronic cigarette) — Participants will be provided with electronic cigarettes and 5% nicotine e-liquid cartridges for 8 weeks and encouraged at in-person and phone assessments to use the electronic cigarette any time they would normally smoke. Participants will be able to choose one of two e-liquid flavors (tobacco, menthol) at baseline.
  Arms: Electronic Cigarette
Other: Nicotine (nicotine pouch) — Participants will be provided with 4mg nicotine pouches for 8 weeks and encouraged at in-person and phone assessments to use the nicotine pouches any time they would normally smoke. Participants will be able to choose one of two nicotine pouch flavors (tobacco, mint) at baseline.
  Arms: Nicotine Pouch

SUMMARY:
This study investigates whether providing 8 weeks of complimentary electronic cigarettes (EC) or nicotine pouches (NP) to low socioeconomic status (SES) adults who smoke and are unable or unwilling to quit smoking will lead to: a) substitution of cigarette smoking with EC or NP; and b) reduced biological indicators of tobacco use and harm relative to those continuing to smoke as usual. This study also examines the feasibility and acceptability of providing EC or NP to help substitution of combustible cigarettes, exploring willingness to participate, continuing with the study, and barriers to substitution through interviews. This project will enroll 45 low SES adults who smoke and will be randomized to one of the three groups that will be followed for 8 weeks: EC, NP, or smoking as usual.

The first study hypothesis is that participants receiving EC or NP will smoke fewer cigarettes per day and have lower cigarette dependence at Week 8 relative to their baseline level, and when compared to the control group. The second hypothesis is that those in the EC or NP group will have greater cigarette abstinence than those smoking as usual at Week 8. There are no anticipated differences between those receiving EC and NP. The third hypothesis is that biological indicators of tobacco use and harm will be lower in those receiving EC or NP relative to their baseline level, and when compared to the control group. The hypothesis is that these biological indicators will be lower in those receiving NP than EC.

DETAILED DESCRIPTION:
This study investigates whether providing 8 weeks of complimentary electronic cigarettes (EC) or nicotine pouches (NP) to low socioeconomic status (SES) adults who smoke and are unable or unwilling to quit smoking will lead to: a) substitution of cigarette smoking with EC or NP; and b) reduced biological indicators of tobacco use and harm relative to those continuing to smoke as usual. This study also examines the feasibility and acceptability of providing EC or NP to help substitution of combustible cigarettes, exploring willingness to participate, continuing with the study, and barriers to substitution through interviews. This project will enroll 45 low SES adults who smoke and will be randomized to one of the three groups that will be followed for 8 weeks: EC, NP, or smoking as usual. At the start of the study, participants will provide informed consent; biological indicators and self-report measures will be collected; and participants will be randomly assigned to one of the 3 groups. Participants in the EC or NP groups will be allowed to experiment with EC or NP flavors prior to receiving an adequate supply of the product to fully substitute combustible smoking for four weeks. Participants in these two groups will also receive encouragement to fully switch from cigarettes to EC or NP. Participants will have 3 in-person visits (baseline, week 4, week 8) and 4 phone visits (weeks 1, 3, 7, and 16). At the week 4 in-person visit, participants will receive a second four-week product supply. Participants will also receive ongoing encouragement to fully substitute with EC or NPs whenever participants would normally smoke. Biomarkers and self-report measures will be reassessed at the Week 8 visit after which participants will complete a debriefing interview. Participants will complete a final report at Week 16.

The first study hypothesis is that participants receiving EC or NP will smoke fewer cigarettes per day and have lower cigarette dependence at Week 8 relative to their baseline level, and when compared to the control group. The second hypothesis is that those in the EC or NP group will have greater cigarette abstinence than those smoking as usual at Week 8. There are no anticipated differences between those receiving EC and NP. The third hypothesis is that biological indicators of tobacco use and harm will be lower in those receiving EC or NP relative to their baseline level, and when compared to the control group. The hypothesis is that these biological indicators will be lower in those receiving NP than EC.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 (inclusive) years of age or greater
2. Past 6 months daily smoking of ≥ 5 cigarettes/day
3. Exhaled CO ≥ 6 ppm at baseline
4. Household income < 250% federal poverty level (FPL)
5. Willingness to substitute combustible cigarettes for EC or NPs
6. Ability to read and write in English
7. Own a telephone (landline or cellphone)

Exclusion Criteria:

1. Intention to quit smoking during the next 30 days
2. Current or past 30 day engagement in smoking cessation
3. Current use of EC or NP ≥ 4 days per month
4. Current self-report of primarily using tobacco products that are not combustible cigarettes
5. Urine-screened pregnancy
6. Hospitalization for a psychiatric issue in the past 30 days or visible instability
7. Other household member is a study participant
8. Participating in another clinical trial at the same time
9. Heart-related event in the past 30 days
10. Planning to move out of the Providence area in the next six months

Note: Cannabis use will be assessed but not excluded

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-02-09 (Estimated)

PRIMARY OUTCOMES:
Change in cigarettes per day from baseline to week 8 | Assessed at baseline and week 8.
  Within and between group difference in past week average cigarettes per day assessed using timeline follow-back (TLFB)
Change in cigarette dependence from baseline to week 8 | Assessed at baseline and week 8.
  Change in cigarette dependence within group and between groups. Assessed using the Strong et al measure adapted from the Population Assessment of Tobacco and Health survey
Cigarette abstinence at week 8 | Week 8.
  Past week any-use of cigarettes assessed using timeline follow-back (TLFB).

SECONDARY OUTCOMES:
Change in Carbon monoxide from baseline to week 8 | Assessed at baseline and week 8.
  Exhaled carbon monoxide assessed via Smokerlyzer and compared within group and between groups.
Change in cotinine from baseline to week 8 | Assessed at baseline and week 8.
  Creatinine-adjusted cotinine assessed via urine compared within group and between groups.
Change in NNAL from baseline to week 8 | Assessed at baseline and week 8.
  4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL), a ratio of NNAL to creatinine-adjusted cotinine assessed via urine and compared within group and between groups.
Change in 8-isoprostane from baseline to week 8 | Assessed at baseline and week 8.
  8-isoprostane assessed via urine and compared within group and between groups
Feasibility and acceptability | through study completion, an average of 6 months
  Willingness to participate as measured by proportion of eligible participants following in-person screening who enroll in the study. Retention as measured by weeks of study participation. Barriers to substitution as indicated in qualitative exit interview.

CONTACTS AND LOCATIONS:
Overall Officials: Jasjit S Ahluwalia, MD, Principal Investigator — Brown University
Locations (1):
- Center for Alcohol and Addiction Studies, Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data except for transcriptions of qualitative interviews will be made available after the completion of all study activities.
Supporting Information: Study Protocol, Analytic Code
Time Frame: After closing the study IRB protocol and destroying all identifiers. Anticipated 2 years after completion of primary data collection. Data availability will be perpetual. Data dissemination plan is pending.

REFERENCES:
- [Derived] Avila JC, Maglalang DD, Nollen NL, Lee SC, Suh R, Malone M, Binjrajka U, Ahluwalia JS. Using Pod Based e-Cigarettes and Nicotine Pouches to Reduce Harm for Adults With Low Socioeconomic Status Who Smoke: A Pilot Randomized Controlled Trial. Nicotine Tob Res. 2024 Aug 22;26(9):1150-1158. doi: 10.1093/ntr/ntae047. PMID 38447095

DOCUMENTS (1):
  • Informed Consent Form (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT05327439/ICF_000.pdf